CLINICAL TRIAL: NCT03865836
Title: Named Patient or Compassionate Use for Treatment Use of ATB200/AT2221 for Patients With Pompe Disease
Brief Title: Expanded Access for ATB200/AT2221 for the Treatment of Pompe Disease
Status: Available | Type: Expanded Access
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ATB200-11
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pompe Disease
Keywords: expanded access; compassionate use
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: ATB200
Drug: AT2221

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to ATB200/AT2221.

DETAILED DESCRIPTION:
This program is being offered on a patient by patient basis and will require company, IRB/IEC and single patient IND approval.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a diagnosis of Pompe disease based on documentation of one of the following:

   1. deficiency of GAA enzyme
   2. GAA genotyping
2. Patient does not currently qualify for an Amicus sponsored on-going clinical trial or is declining on currently approved ERT (e.g. Myozyme)
3. The patient must be willing to receive treatment with ATB200/AT2221 via this program, which includes signing an authorization form for sharing clinical data with Amicus Therapeutics, and its agent Early Access Care LLC.

Exclusion Criteria:

1. Patient, whether male or female, is planning to conceive a child during the treatment program.
2. Patient has a hypersensitivity to any of the excipients in ATB200, alglucosidase alfa, or AT2221
3. Patient has a medical or any other extenuating condition or circumstance that may, in the opinion of the investigator, pose an undue safety risk to the subject or compromise his/her ability to comply with or adversely impact protocol requirements.
4. Patient has received any gene therapy at any time.
5. Concomitant use of miglitol (eg, Glyset), non-AT2221 form of miglustat (eg, Zavesca), acarbose (eg, Precose or Glucobay), voglibose (eg, Volix, Vocarb, or Volibo)

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Related Info — https://clinicaltrials.gov/ct2/show/NCT03729362?term=ATB200-03&rank=1